CLINICAL TRIAL: NCT03112395
Title: Local Application of Combined Optical and Magnetic Stimulation (COMS) in Patients Suffering From Chronic Wounds at Lower Extremities: Safety Evaluation
Brief Title: Local Application of Combined Optical and Magnetic Stimulation (COMS) for Treatment of Chronic Wounds: Safety Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piomic Medical AG (Industry)
Collaborators: Venenklinik Bellevue (Other); Kantonsspital Nidwalden (Unknown); Spital Männedorf (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMS_01
Record Dates: First submitted 2017-04-03; First posted 2017-04-13 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2019-10

CONDITIONS: Leg Ulcers Venous; Leg Ulcer Arterial; Leg Ulcer Mixed
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined SOC/Pio treatment (Experimental): Prospective trial (1 month SOC, 2 month SOC + Pio Medical Device, 1 month SOC follow-up) month, with collection of endpoints every second week
  Interventions: Device: Pio Medical Device

INTERVENTIONS:
Device: Pio Medical Device — The Pio device combines the technologies of pulse modulated magnetic fields and light emission locally applied to the wound area.

SUMMARY:
The demographic shift and the increasing prevalence of chronic wounds represent major challenges for modern health care systems. Classic chronic wounds (venous ulcer, arterial ulcer, mixed ulcer) persist for months or years with a very slow or even no healing progress. Patients suffer from pain and immobility, which dramatically reduces their quality of life. Complications such as infections or tissue necrosis can lead to a bad outcome and amputation of extremities.

The Pio device offers a non-invasive and non-toxic therapeutic approach. The system combines the technologies of pulse modulated magnetic fields and light emission locally applied to the wound area. The investigational medical device represents a promising combinational therapeutic approach to synergistically increase the tissues regenerative potential. By stimulating electrophysiological processes at the site of injury, the cells regain its capacity to efficiently regenerate the injured or diseased tissue. It is expected that the patient benefits from a faster healing process, reduced inflammation as well as an improved overall treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Male and female patients
* Age: 18 - 90
* Chronic wound (venous ulcer, arterial ulcer, mixed ulcer) since at least 4 weeks
* Wound area minimal 1 cm2, maximal 50 cm2
* No adaptions for treatment of causal therapy of disease

Exclusion Criteria:

* Women who are pregnant
* Known or suspected non-compliance, drug or alcohol abuse,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Patients with active devices (e.g. Pacemakers and defibrillators, infusion devices, insulin pumps)
* Metallic implants and endoprosthesis at extremities lower than hip
* Life threatening condition
* Immunosuppressive after foreign organ transplant or chemotherapeutic treatment within 30 days before study begin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event | At each visit, up to 16 weeks
  The incidence of adverse events will be assessed at each visit, prior to the Pio treatment and directly after the Pio treatment. The incidence of treatment-emergent adverse events will be compared to the incidence of standard of care emergent adverse events.
Severity of adverse event | At each visit, up to 16 weeks
  The severity of adverse events will be assessed at each visit, prior to the Pio treatment and directly after the Pio treatment. The severity of treatment-emergent adverse events will be compared to the severity of standard of care emergent adverse events.
Time of occurrence of adverse event | At each visit, up to 16 weeks
  The time of occurrence of adverse events will be assessed at each visit, prior to the Pio treatment and directly after the Pio treatment. The time of occurrence of treatment-emergent adverse events will be compared to the time of occurrence of standard of care emergent adverse events.
Type of adverse event | At each visit, up to 16 weeks
  The type of adverse events will be assessed at each visit, prior to the Pio treatment and directly after the Pio treatment. The type of treatment-emergent adverse events will be compared to the type of standard of care emergent adverse events.

SECONDARY OUTCOMES:
Wound area | At first visit of the week, before Pio treatment, up to 16 weeks
  The wound area will be measured weekly right before the Pio treatment.
Wound volume | At first visit of the week, before Pio treatment, up to 16 weeks
  The wound volume will be measured weekly right before the Pio treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Traber, Dr. med, Principal Investigator — Venenklinik Bellevue; Christiane Bittner, Dr. med., Principal Investigator — Kantonsspital Nidwalden; Georg Liesch, Dr. med, Principal Investigator — Spital Männedorf
Locations (3):
- Switzerland (3):
  - Kantonsspital Nidwalden, Stans, Ennetmooserstrasse 19
  - Venenklinik Bellevue, Kreuzlingen
  - Spital Männedorf, Zurich